CLINICAL TRIAL: NCT03145649
Title: Breast Milk Hormones and Early Infant Growth of Women With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D111100000611001
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gestational Diabetes
Keywords: Breast milk; Hormone; Infant growth; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk specimens were collected from women during lactation period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes mellitus: Women with gestational diabetes mellitus and their infants. The blood glucose of women with gestational diabetes mellitus was controlled by dietary therapy or insulin injection.
  Interventions: Other: Dietary therapy or insulin injection
- Healthy: Healthy mother-infant dyads

INTERVENTIONS:
Other: Dietary therapy or insulin injection
  Groups: Gestational diabetes mellitus

SUMMARY:
Background: Breastfeeding has been associated with attenuated risk of obesity and type 2 diabetes in children born to women with diabetes. However, breast milk (BM) components responsible for the protective effects remain to be unveiled.

Objective: To evaluate the hormone concentrations in BM of women with gestational diabetes mellitus (GDM) and their influence on early infant growth.

Design: The investigators followed nulliparous women with and without GDM and their breastfed term singletons. Women diagnosed with GDM received dietary therapy or insulin injection to maintain euglycemia during pregnancy. Hormone concentrations in BM (i.e., adiponectin, leptin, insulin, and ghrelin) were tested and infant growth was evaluated on days 3, 42 and 90. The investigators compared the hormone concentrations between the GDM and healthy groups, and tested the associations of hormone concentrations with maternal factors (i.e., BMI, plasma glucose concentration, gestational age, and delivery mode) and early infant growth.

Hypothesis: Hormone concentrations in BM could be determined by multiple maternal factors, including metabolic and obstetrical factors. GDM should be a significant influencing factor for hormone concentrations in BM.

DETAILED DESCRIPTION:
Subjects Nulliparous women with GDM and healthy women, who intended to exclusively breastfeed their singletons, were recruited consecutively from the obstetric wards at the Peking Union Medical College Hospital and the Beijing Obstetrics and Gynecology Hospital during the 37th gestational week. The exclusion criteria were: pre-pregnancy diabetes, fetal anomaly, gestational hypertension, preeclampsia, fetal growth restriction, ruptured membranes, postpartum glucose abnormalities (see below), and introduction of formula feeding during the follow-ups. Women with plasma glucose>7.8mmol/L in the 1-hour 50g glucose load test (GLT) during the 24th-28th gestational weeks underwent a 3-hour 100g diagnostic oral glucose tolerance test (OGTT) following a 12-hour overnight fast. GDM was diagnosed if two or more plasma glucose reads in the OGTT equaled or exceeded the threshold according to Carpenter and Coustan. All subjects diagnosed with GDM initially received dietary therapy to attain glycemic targets: 3.3-5.6 mmol/L at fasting, 3.3-5.8 mmol/L pre-prandially, 4.4-6.7 mmol/L 2-hours post-prandially, and 4.4-6.7 mmol/L at night. The participants were followed by dietitians to ensure euglycemia, appropriate weight gain, and adequate nutritional intake. The participants who did not attain glycemic targets in 2 weeks after starting the dietary therapy were given insulin via injection. As macronutrients in BM were mainly determined by the maternal glucose metabolic status, the investigators excluded women with postpartum glucose abnormalities, i.e., impaired glucose tolerance (IGT) with the 2-hour plasma glucose between 7.8 and 11.0 mmol/l and type 2 diabetes with the 2-hour plasma glucose ≥11.1 mmol/l in the 75g OGTT on postpartum day 42.

Anthropometric measurements Data was recorded using customized case report forms. Obstetric data, such as glycemic tests, gestational age, and mode of delivery, were retrieved from the medical records. Pre-pregnancy weight was self-reported. Mothers' height was measured twice to the nearest 0.1 cm with a wall-mounted stadiometer. Mothers' weight was measured twice to the nearest 0.1 kg with a medical balance scale before delivery, on postpartum days 42 and 90. The weight, length, and head circumference of the infants were measured at birth, on days 42 and 90. The infants were weighed twice in nude using a precision scale (Seca, CA, USA). Body length and head circumference were measured twice to the nearest 0.1 cm with a length board and non-stretchable measuring tapes (Seca, CA, USA). The mean values of the two readings were used for data analysis.

Milk sample collection, processing, and laboratory tests Colostrum samples were collected between 8 a.m. and 9 a.m. before infant feeding on the third day after delivery. Mature milk, including both foremilk and hindmilk, was delivered and collected from one breast before infant feeding using an electric pump (Medela, Baar, Switzerland) between 2 p.m. and 4 p.m. on days 42 and 90 in the clinics. The milk samples were frozen immediately in sterilized plastic tubes at -80°C. Before quantifying the hormones in BM, the samples were thawed at 4°C, sonicated, and centrifuged. The samples were sonicated using a sonicator (Braun-sonic sonicator, B. Braun, Melsungen, Germany) at 50 watts for 3 bursts with 10-second intervals, and centrifuged at 100,000g for 1 hour at 4°C. The supernatant fat was discarded and the skim milk was used for quantifying adiponectin, leptin, insulin, and ghrelin by ELISA at the Key Laboratory of Endocrinology in the Peking Union Medical College Hospital. The assay had an intra- and inter-assay CV of <5.4 and <8.5% for adiponectin, and <7.4% and <9.3% for leptin, respectively. The insulin assay had no cross-reactivity to proinsulin (<0.05%), and had sensitivity of 0.5 mU/L and an inter-assay CV of <9.0%. Total ghrelin was tested using the total human ghrelin ELISA kit (Millipore, USA). The intra- and inter-assay CVs for the ghrelin assay were <1.9% and <7.7%.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women with GDM and healthy women, who intended to exclusively breastfeed their singletons, were recruited consecutively from the obstetric wards at the Peking Union Medical College Hospital and the Beijing Obstetrics and Gynecology Hospital during the 37th gestational week.

Exclusion Criteria:

* Pre-pregnancy diabetes, fetal anomaly, gestational hypertension, preeclampsia, fetal growth restriction, ruptured membranes, postpartum glucose abnormalities, and introduction of formula feeding during the follow-ups.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects were recruited consecutively from the obstetric wards at the Peking Union Medical College Hospital and the Beijing Obstetrics and Gynecology Hospital.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2010-10-21 (Actual); Study Completion 2011-07-16 (Actual)

PRIMARY OUTCOMES:
Adiponectin in the colostrum | Day 3 after delivery
  Adiponectin concentration in the colostrum
Leptin in the colostrum | Day 3 after delivery
  Leptin concentration in the colostrum
Insulin in the colostrum | Day 3 after delivery
  Insulin concentration in the colostrum
Ghrelin in the colostrum | Day 3 after delivery
  Ghrelin concentration in the colostrum
Adiponectin in the early mature milk | Day 42 after delivery
  Adiponectin concentration in the mature milk of day 42
Leptin in the early mature milk | Day 42 after delivery
  Leptin concentration in the mature milk of day 42
Insulin in the early mature milk | Day 42 after delivery
  Insulin concentration in the mature milk of day 42
Ghrelin in the early mature milk | Day 42 after delivery
  Ghrelin concentration in the mature milk of day 42
Adiponectin in the mature milk | Day 90 after delivery
  Adiponectin concentration in the mature milk of day 90
Leptin in the mature milk | Day 90 after delivery
  Leptin concentration in the mature milk of day 90
Insulin in the mature milk | Day 90 after delivery
  Insulin concentration in the mature milk of day 90
Ghrelin in the mature milk | Day 90 after delivery
  Ghrelin concentration in the mature milk of day 90
Infant birth weight | At birth
  Infants' weight at birth
Infant birth height | At birth
  Infants' height at birth
Infant birth head circumference | At birth
  Infants' head circumference at birth
Infant weight at day 42 | Day 42
  Infants' weight at day 42
Infant height at day 42 | Day 42
  Infants' height at day 42
Infant head circumference at day 42 | Day 42
  Infants' head circumference at day 42
Infant weight at day 90 | Day 90
  Infants' weight at day 90
Infant height at day 90 | Day 90
  Infants' height at day 90
Infant head circumference at day 90 | Day 90
  Infants' head circumference at day 90

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dosch HM, Becker DJ. Infant feeding and autoimmune diabetes. Adv Exp Med Biol. 2002;503:133-40. doi: 10.1007/978-1-4615-0559-4_15. No abstract available. PMID 12026012
- [Background] Catalano PM, McIntyre HD, Cruickshank JK, McCance DR, Dyer AR, Metzger BE, Lowe LP, Trimble ER, Coustan DR, Hadden DR, Persson B, Hod M, Oats JJ; HAPO Study Cooperative Research Group. The hyperglycemia and adverse pregnancy outcome study: associations of GDM and obesity with pregnancy outcomes. Diabetes Care. 2012 Apr;35(4):780-6. doi: 10.2337/dc11-1790. Epub 2012 Feb 22. PMID 22357187
- [Background] Logan KM, Emsley RJ, Jeffries S, Andrzejewska I, Hyde MJ, Gale C, Chappell K, Mandalia S, Santhakumaran S, Parkinson JR, Mills L, Modi N. Development of Early Adiposity in Infants of Mothers With Gestational Diabetes Mellitus. Diabetes Care. 2016 Jun;39(6):1045-51. doi: 10.2337/dc16-0030. Epub 2016 May 12. PMID 27208326
- [Background] Gillman MW, Rifas-Shiman S, Berkey CS, Field AE, Colditz GA. Maternal gestational diabetes, birth weight, and adolescent obesity. Pediatrics. 2003 Mar;111(3):e221-6. doi: 10.1542/peds.111.3.e221. PMID 12612275
- [Background] Sellers EA, Dean HJ, Shafer LA, Martens PJ, Phillips-Beck W, Heaman M, Prior HJ, Dart AB, McGavock J, Morris M, Torshizi AA, Ludwig S, Shen GX. Exposure to Gestational Diabetes Mellitus: Impact on the Development of Early-Onset Type 2 Diabetes in Canadian First Nations and Non-First Nations Offspring. Diabetes Care. 2016 Dec;39(12):2240-2246. doi: 10.2337/dc16-1148. Epub 2016 Oct 4. PMID 27703026
- [Background] Houseknecht KL, McGuire MK, Portocarrero CP, McGuire MA, Beerman K. Leptin is present in human milk and is related to maternal plasma leptin concentration and adiposity. Biochem Biophys Res Commun. 1997 Nov 26;240(3):742-7. doi: 10.1006/bbrc.1997.7736. PMID 9398637
- [Background] Weyermann M, Beermann C, Brenner H, Rothenbacher D. Adiponectin and leptin in maternal serum, cord blood, and breast milk. Clin Chem. 2006 Nov;52(11):2095-102. doi: 10.1373/clinchem.2006.071019. Epub 2006 Sep 21. PMID 16990422
- [Background] Savino F, Lupica MM, Benetti S, Petrucci E, Liguori SA, Cordero Di Montezemolo L. Adiponectin in breast milk: relation to serum adiponectin concentration in lactating mothers and their infants. Acta Paediatr. 2012 Oct;101(10):1058-62. doi: 10.1111/j.1651-2227.2012.02744.x. Epub 2012 Jul 12. PMID 22646778
- [Background] Bronsky J, Mitrova K, Nevoral J, Zamecnik J. Immunoexpression of type-1 adiponectin receptor in the human intestine. Cesk Patol. 2012 Jul;48(3):165-6. PMID 23057433
- [Background] Hansen GH, Niels-Christiansen LL, Danielsen EM. Leptin and the obesity receptor (OB-R) in the small intestine and colon: a colocalization study. J Histochem Cytochem. 2008 Jul;56(7):677-85. doi: 10.1369/jhc.2008.950782. Epub 2008 Apr 14. PMID 18413648
- [Background] Georgiev IP, Georgieva TM, Pfaffl M, Hammon HM, Blum JW. Insulin-like growth factor and insulin receptors in intestinal mucosa of neonatal calves. J Endocrinol. 2003 Jan;176(1):121-32. doi: 10.1677/joe.0.1760121. PMID 12525256
- [Background] Mitrovic O, Cokic V, Dikic D, Budec M, Vignjevic S, Suboticki T, Diklic M, Ajtic R. Ghrelin receptors in human gastrointestinal tract during prenatal and early postnatal development. Peptides. 2014 Jul;57:1-11. doi: 10.1016/j.peptides.2014.04.010. Epub 2014 Apr 23. PMID 24768902
- [Background] Correa A, Bardenheier B, Elixhauser A, Geiss LS, Gregg E. Trends in prevalence of diabetes among delivery hospitalizations, United States, 1993-2009. Matern Child Health J. 2015 Mar;19(3):635-42. doi: 10.1007/s10995-014-1553-5. PMID 24996952
- [Background] Chamberlain C, Banks E, Joshy G, Diouf I, Oats JJ, Gubhaju L, Eades S. Prevalence of gestational diabetes mellitus among Indigenous women and comparison with non-Indigenous Australian women: 1990-2009. Aust N Z J Obstet Gynaecol. 2014 Oct;54(5):433-40. doi: 10.1111/ajo.12213. Epub 2014 Apr 29. PMID 24773552
- [Background] van Beusekom CM, Zeegers TA, Martini IA, Velvis HJ, Visser GH, van Doormaal JJ, Muskiet FA. Milk of patients with tightly controlled insulin-dependent diabetes mellitus has normal macronutrient and fatty acid composition. Am J Clin Nutr. 1993 Jun;57(6):938-43. doi: 10.1093/ajcn/57.6.938. PMID 8503365
- [Result] Schack-Nielsen L, Michaelsen KF. Breast feeding and future health. Curr Opin Clin Nutr Metab Care. 2006 May;9(3):289-96. doi: 10.1097/01.mco.0000222114.84159.79. PMID 16607131
- [Result] Armstrong J, Reilly JJ; Child Health Information Team. Breastfeeding and lowering the risk of childhood obesity. Lancet. 2002 Jun 8;359(9322):2003-4. doi: 10.1016/S0140-6736(02)08837-2. PMID 12076560
- [Result] Owen CG, Martin RM, Whincup PH, Smith GD, Cook DG. Does breastfeeding influence risk of type 2 diabetes in later life? A quantitative analysis of published evidence. Am J Clin Nutr. 2006 Nov;84(5):1043-54. doi: 10.1093/ajcn/84.5.1043. PMID 17093156
- [Result] Crume TL, Ogden L, Maligie M, Sheffield S, Bischoff KJ, McDuffie R, Daniels S, Hamman RF, Norris JM, Dabelea D. Long-term impact of neonatal breastfeeding on childhood adiposity and fat distribution among children exposed to diabetes in utero. Diabetes Care. 2011 Mar;34(3):641-5. doi: 10.2337/dc10-1716. PMID 21357361
- [Result] Crume TL, Ogden LG, Mayer-Davis EJ, Hamman RF, Norris JM, Bischoff KJ, McDuffie R, Dabelea D. The impact of neonatal breast-feeding on growth trajectories of youth exposed and unexposed to diabetes in utero: the EPOCH Study. Int J Obes (Lond). 2012 Apr;36(4):529-34. doi: 10.1038/ijo.2011.254. Epub 2012 Jan 31. PMID 22290537
- [Result] Savino F, Benetti S, Liguori SA, Sorrenti M, Cordero Di Montezemolo L. Advances on human milk hormones and protection against obesity. Cell Mol Biol (Noisy-le-grand). 2013 Nov 3;59(1):89-98. PMID 24200024
- [Result] Shehadeh N, Khaesh-Goldberg E, Shamir R, Perlman R, Sujov P, Tamir A, Makhoul IR. Insulin in human milk: postpartum changes and effect of gestational age. Arch Dis Child Fetal Neonatal Ed. 2003 May;88(3):F214-6. doi: 10.1136/fn.88.3.f214. PMID 12719395
- [Result] Martin LJ, Woo JG, Geraghty SR, Altaye M, Davidson BS, Banach W, Dolan LM, Ruiz-Palacios GM, Morrow AL. Adiponectin is present in human milk and is associated with maternal factors. Am J Clin Nutr. 2006 May;83(5):1106-11. doi: 10.1093/ajcn/83.5.1106. PMID 16685053
- [Result] Schuster S, Hechler C, Gebauer C, Kiess W, Kratzsch J. Leptin in maternal serum and breast milk: association with infants' body weight gain in a longitudinal study over 6 months of lactation. Pediatr Res. 2011 Dec;70(6):633-7. doi: 10.1203/PDR.0b013e31823214ea. PMID 21857386
- [Result] Andreas NJ, Hyde MJ, Gale C, Parkinson JR, Jeffries S, Holmes E, Modi N. Effect of maternal body mass index on hormones in breast milk: a systematic review. PLoS One. 2014 Dec 23;9(12):e115043. doi: 10.1371/journal.pone.0115043. eCollection 2014. PMID 25536196
- [Result] Dundar NO, Dundar B, Cesur G, Yilmaz N, Sutcu R, Ozguner F. Ghrelin and adiponectin levels in colostrum, cord blood and maternal serum. Pediatr Int. 2010 Aug;52(4):622-5. doi: 10.1111/j.1442-200X.2010.03100.x. PMID 20202158
- [Result] Fields DA, Demerath EW. Relationship of insulin, glucose, leptin, IL-6 and TNF-alpha in human breast milk with infant growth and body composition. Pediatr Obes. 2012 Aug;7(4):304-12. doi: 10.1111/j.2047-6310.2012.00059.x. Epub 2012 May 10. PMID 22577092
- [Result] Aydin S, Geckil H, Karatas F, Donder E, Kumru S, Kavak EC, Colak R, Ozkan Y, Sahin I. Milk and blood ghrelin level in diabetics. Nutrition. 2007 Nov-Dec;23(11-12):807-11. doi: 10.1016/j.nut.2007.08.015. PMID 17936195
- [Result] Aydin S. The presence of the peptides apelin, ghrelin and nesfatin-1 in the human breast milk, and the lowering of their levels in patients with gestational diabetes mellitus. Peptides. 2010 Dec;31(12):2236-40. doi: 10.1016/j.peptides.2010.08.021. Epub 2010 Sep 8. PMID 20813143
- [Result] Ley SH, Hanley AJ, Sermer M, Zinman B, O'Connor DL. Associations of prenatal metabolic abnormalities with insulin and adiponectin concentrations in human milk. Am J Clin Nutr. 2012 Apr;95(4):867-74. doi: 10.3945/ajcn.111.028431. Epub 2012 Feb 29. PMID 22378730
- [Result] Woo JG, Guerrero ML, Altaye M, Ruiz-Palacios GM, Martin LJ, Dubert-Ferrandon A, Newburg DS, Morrow AL. Human milk adiponectin is associated with infant growth in two independent cohorts. Breastfeed Med. 2009 Jun;4(2):101-9. doi: 10.1089/bfm.2008.0137. PMID 19500050
- [Result] Woo JG, Guerrero ML, Guo F, Martin LJ, Davidson BS, Ortega H, Ruiz-Palacios GM, Morrow AL. Human milk adiponectin affects infant weight trajectory during the second year of life. J Pediatr Gastroenterol Nutr. 2012 Apr;54(4):532-9. doi: 10.1097/MPG.0b013e31823fde04. PMID 22094897
- [Result] Cesur G, Ozguner F, Yilmaz N, Dundar B. The relationship between ghrelin and adiponectin levels in breast milk and infant serum and growth of infants during early postnatal life. J Physiol Sci. 2012 May;62(3):185-90. doi: 10.1007/s12576-012-0193-z. Epub 2012 Feb 5. PMID 22311236
- [Result] Doneray H, Orbak Z, Yildiz L. The relationship between breast milk leptin and neonatal weight gain. Acta Paediatr. 2009 Apr;98(4):643-7. doi: 10.1111/j.1651-2227.2008.01192.x. Epub 2009 Jan 7. PMID 19141141
- [Result] Savino F, Fissore MF, Liguori SA, Oggero R. Can hormones contained in mothers' milk account for the beneficial effect of breast-feeding on obesity in children? Clin Endocrinol (Oxf). 2009 Dec;71(6):757-65. doi: 10.1111/j.1365-2265.2009.03585.x. Epub 2009 Mar 19. PMID 19302580
- [Result] Weyermann M, Brenner H, Rothenbacher D. Adipokines in human milk and risk of overweight in early childhood: a prospective cohort study. Epidemiology. 2007 Nov;18(6):722-9. doi: 10.1097/ede.0b013e3181567ed4. PMID 18062063